CLINICAL TRIAL: NCT00282308
Title: A Phase II, Randomized, Parallel-group, Open-label, Multicenter Study to Evaluate the Effects of Rituximab on Immune Responses in Subjects With Active Rheumatoid Arthritis Receiving Background Methotrexate
Brief Title: A Study to Evaluate the Effects of Rituximab on Immune Responses in Subjects With Active Rheumatoid Arthritis Receiving Background Methotrexate
Acronym: SIERRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U3374g
Record Dates: First submitted 2006-01-24; First posted 2006-01-26 (Estimated); Results first posted 2013-10-21 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-07

CONDITIONS: Rheumatoid Arthritis
Keywords: RA; Rituxan; SIERRA
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab; Methotrexate; 23-valent pneumococcal capsular polysaccharide vaccine; keyhole-limpet hemocyanin

ARMS (2):
- Rituximab + methotrexate (Group A) (Experimental): Patients received 2 intravenous infusions of rituximab 1000 mg, 14 days apart + methotrexate 10-25 mg/wk orally or subcutaneously during the Treatment Period.
  Interventions: Drug: Rituximab; Drug: Methotrexate; Drug: Methylprednisone; Biological: C. albicans; Biological: Tetanus toxoid adsorbed booster vaccine; Biological: 23-valent pneumococcal polysaccharide vaccine; Biological: Keyhole limpet hemocyanin
- Methotrexate (Group B) (Active Comparator): Patients received methotrexate 10-25 mg/wk orally or subcutaneously during the Treatment Period.
  Interventions: Drug: Methotrexate; Biological: C. albicans; Biological: Tetanus toxoid adsorbed booster vaccine; Biological: 23-valent pneumococcal polysaccharide vaccine; Biological: Keyhole limpet hemocyanin

INTERVENTIONS:
Drug: Rituximab — Rituximab was supplied in single-use vials.
  Other Names: Rituxan; MabThera
  Arms: Rituximab + methotrexate (Group A)
Drug: Methotrexate
Drug: Methylprednisone — Patients received methylprednisolone 100 mg intravenously before each infusion of rituximab.
  Arms: Rituximab + methotrexate (Group A)
Biological: C. albicans — Patients received an intradermal injection of C. albicans (0.1 mL) on the volar surface of the forearm.
Biological: Tetanus toxoid adsorbed booster vaccine — Patients received an intramuscular injection of the tetanus toxoid adsorbed booster vaccine (1 mg in 0.5 mL) in the deltoid muscle.
Biological: 23-valent pneumococcal polysaccharide vaccine — Patients received an intramuscular injection of the 23-valent pneumococcal polysaccharide vaccine (0.5 mL) in the deltoid muscle.
Biological: Keyhole limpet hemocyanin — Patients received a subcutaneous injection of keyhole limpet hemocyanin (1 mg)

SUMMARY:
This was a Phase II, randomized, open-label, multicenter study designed to evaluate the immune response to vaccines after administration of 1000 mg of rituximab in subjects with active rheumatoid arthritis (RA) who were receiving background methotrexate (MTX).

DETAILED DESCRIPTION:
Patients were randomized to 2 groups in this study: Group A (active group) and Group B (control group). Patients with active rheumatic arthritis treated with rituximab in combination with methotrexate (Group A) were compared with patients treated with methotrexate alone (Group B).

Group A

Group A patients received rituximab 1000 mg intravenously (IV) on Days 3 and 17 of the 36 week treatment period.

At Day 1 and at Week 24, patients received an intradermal injection of 0.1 mL of C. albicans on the volar surface of the forearm. Forty-eight to 72 hours after each injection, patients were evaluated for a delayed-type hypersensitivity response by measuring the diameter of induration (palpable raised, hardened area of the forearm skin).

At Week 24, patients received a tetanus toxoid adsorbed booster vaccine (1 mg in 0.5 mL) intramuscular (IM) injection in the deltoid muscle. Serum levels of tetanus toxoid titers were obtained at Day 3 immediately prior to the first administration of rituximab, and immediately prior to and 4 weeks after administration of the tetanus toxoid adsorbed vaccine.

At Week 28, patients received an IM injection of the 23-valent pneumococcal polysaccharide vaccine (0.5 mL) in the deltoid muscle. Serum levels for antibodies to 12 pneumococcal serotypes were measured at Day 3 immediately prior to the first administration of rituximab, and immediately prior to and 4 weeks after administration of the pneumococcal vaccine.

At Weeks 32 and 33, patients received subcutaneous (SC) keyhole limpet hemocyanin 1 mg. Serum anti-keyhole limpet hemocyanin antibody levels were measured at Day 3 immediately prior to the first administration of rituximab, and immediately prior to and 4 weeks after the first administration of keyhole limpet hemocyanin.

Samples were obtained for the determination of serum rituximab concentration (pharmacokinetics), peripheral blood CD19 counts (pharmacodynamics), and the presence of human anti-chimeric antibodies from all patients in Group A.

Group A patients completed the treatment period at Week 36 and, if qualified, had the option of entering the optional extension re-treatment period. Patients who did not qualify for or who did not choose to receive the optional extension re-treatment entered the approximately 1-year safety follow-up period. After the safety follow-up period, patients who remained peripherally CD19-positive B-cell depleted entered the B-cell follow-up period where they were followed every 12 weeks until their peripheral CD19-positive B cells returned to baseline values or the lower limit of normal, whichever was lower.

Group B

Because the immune response to vaccines was not likely to be influenced by the knowledge of treatment assignment or the time-of-year administration, vaccinations of Group B patients were administered sooner than in the Group A 36 week treatment period.

At Day 1 and at Week 12, patients received an intradermal injection of 0.1 mL of C. albicans on the volar surface of the forearm. Forty-eight to 72 hours after each injection, patients were evaluated for a delayed-type hypersensitivity response by measuring the diameter of induration (palpable raised, hardened area of the forearm skin).

On Day 1, patients received a tetanus toxoid adsorbed booster vaccine (1 mg in 0.5 mL) IM injection in the deltoid muscle. Serum levels of tetanus toxoid titers were obtained immediately prior to and 4 weeks after administration of the tetanus toxoid adsorbed vaccine.

At Week 4, patients received an IM injection of the 23-valent pneumococcal polysaccharide vaccine (0.5 mL) in the deltoid muscle. Serum levels for antibodies to 12 pneumococcal serotypes were measured at Day 1, and immediately prior to and 4 weeks after administration of the pneumococcal vaccine.

At Weeks 8 and 9, patients received SC keyhole limpet hemocyanin 1 mg. Serum anti-keyhole limpet hemocyanin antibody levels were measured at Day 1, and immediately prior to and 4 weeks after the first administration of keyhole limpet hemocyanin.

Upon completion of the Week 12 visit, Group B patients with active rheumatic arthritis, defined as a swollen joint count (SJC) ≥ 4 (66 joint count) and a tender joint count (TJC) ≥ 6 (68 joint count) were eligible for treatment with 2 infusions of rituximab 1000 mg IV, 14 days apart. Patients received the first infusion of rituximab within 2 weeks after completing the Week 12 visit and after the second C. albicans skin test had been read. Patients received methylprednisolone 100 mg IV before each infusion of rituximab.

Group B patients who received treatment with rituximab completed the treatment period through Week 36 and, if qualified, had the option of entering the optional extension re-treatment period. Patients who did not qualify for or who did not choose to receive the optional extension re-treatment entered the approximately 1-year safety follow-up period. After the safety follow-up period, patients who remained peripherally CD19-positive B-cell depleted entered the B-cell follow-up period where they were followed every 12 weeks until their peripheral CD19-positive B cells returned to baseline values or the lower limit of normal, whichever was lower.

Group B patients who did not qualify for and/or did not choose treatment with rituximab completed the study at the end of the primary study period (Week 12).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years.
* Diagnosis of rheumatoid arthritis (RA) for at least 6 months.
* Receiving treatment for RA on an outpatient basis.
* Use of methotrexate (MTX) at a dose of 10-25 mg/wk (oral [PO] or subcutaneous [SC]) for at least 12 weeks prior to Day 1, with the dose stable during the last 4 weeks prior to Day 1 (first day of the treatment period).
* If taking a background corticosteroid, use of the corticosteroid must be for at least 12 weeks prior to Day 1 at a stable dose during the last 4 weeks prior to Day 1.
* If taking one non-steroidal anti-inflammatory drug (NSAID), use of a stable dose for at least 2 weeks prior to Day 1.

Exclusion Criteria:

* Rheumatic autoimmune disease other than RA or significant systemic involvement secondary to RA; Sjogren's syndrome with RA is permitted.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2006-01-23 (Actual); Primary Completion 2008-01-31 (Actual); Study Completion 2012-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariella Kelman, M.D., Study Director — Genentech, Inc.
Locations (34):
- United States (34):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Arthritis & Rheumatology Research, Pllc, Paradise Valley, Arizona
  - Sun Valley Arthritis Center, Peoria, Arizona
  - Desert Medical Advances, Palm Desert, California
  - Inland Rheumatology; Clinical Trials, Inc., Upland, California
  - Arthritis Associates of South Florida, Delray Beach, Florida
  - The Arthritis Center, Palm Harbor, Florida
  - Center For Arthritis; Research Dept, South Miami, Florida
  - Intermountain Orthopaedics, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - Univ of Chicago, Chicago, Illinois
  - Evanston Northwestern Healthcare, Evanston, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Kentuckiana Center For Better Bone & Joint Healthx, Louisville, Kentucky
  - Clinical Research Network, Slidell, Louisiana
  - Johns Hopkins University; Rheumatology, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Rheumatology, P.C.; Medical Arts Building, Kalamazoo, Michigan
  - Borgess Research Institute, Kalamazoo, Michigan
  - Justus Fiechtner MD - PP, Lansing, Michigan
  - Center for Rheumatology, State Uni. of New York, Albany, New York
  - Aair Research Center, Rochester, New York
  - University of Rochester - Strong Memorial Hospital, Rochester, New York
  - Physicians East Pa, Greenville, North Carolina
  - Health Research of Oklahoma, Llc, Oklahoma City, Oklahoma
  - Oregon Health Sciences Uni, Portland, Oregon
  - Altoona Arthritis & Osteo Center, Duncansville, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Rheumatology Associates, Charleston, South Carolina
  - Medical University of S. Carolina, Charleston, South Carolina
  - Arthritis Associates, Hixson, Tennessee
  - Arthritis Care & Diagnostic Center, Dallas, Texas
  - Arthritis Clinic of Northern Virginia, Arlington, Virginia
  - Arthritis Northwest, Spokane, Spokane, Washington

REFERENCES:
- [Derived] Bingham CO 3rd, Looney RJ, Deodhar A, Halsey N, Greenwald M, Codding C, Trzaskoma B, Martin F, Agarwal S, Kelman A. Immunization responses in rheumatoid arthritis patients treated with rituximab: results from a controlled clinical trial. Arthritis Rheum. 2010 Jan;62(1):64-74. doi: 10.1002/art.25034. PMID 20039397

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients (Combined Groups A and B): Patients who qualified for re-treatment received 2 intravenous infusions of rituximab 1000 mg, 14 days apart + methotrexate 10-25 mg/week orally or subcutaneously. Patients received methylprednisolone 100 mg intravenously before each infusion of rituximab. Patients received no treatment during the Safety Follow-up Period.
Period: Treatment Period
Arm/Group | Rituximab + Methotrexate (Group A) | Methotrexate (Group B) | All Patients (Combined Groups A and B)
Started | 69 | 34 | 0 (Participant Flow is reported separately for the treatment groups for this Period.)
Completed | 65 | 28 | 0
Not Completed | 4 | 6 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Subject/Guardian Decision to Withdraw | 2 | 4 | 0
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Not Treated with Study Drug | 1 | 0 | 0
Period: Optional Extension Re-treatment Period
Arm/Group | Rituximab + Methotrexate (Group A) | Methotrexate (Group B) | All Patients (Combined Groups A and B)
Started | 0 (Participant Flow is reported for the combined treatment groups for this Period.) | 0 (Participant Flow is reported for the combined treatment groups for this Period.) | 78 (Not all patients who completed the Treatment Period entered this Optional Re-treatment Period.)
Completed | 0 | 0 | 72
Not Completed | 0 | 0 | 6
Not completed — Adverse Event | 0 | 0 | 4
Not completed — Physician's Decision to Withdraw | 0 | 0 | 1
Not completed — Subject/Guardian Decision to Withdraw | 0 | 0 | 1
Period: Safety Follow-up Period
Arm/Group | Rituximab + Methotrexate (Group A) | Methotrexate (Group B) | All Patients (Combined Groups A and B)
Started | 0 (Participant Flow is reported for the combined treatment groups for this Period.) | 0 (Participant Flow is reported for the combined treatment groups for this Period.) | 100 (Some patients entered this Safety Follow-up Period directly from the Treatment Period.)
Completed | 0 | 0 | 81
Not Completed | 0 | 0 | 19
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 5
Not completed — Physician Decision to Withdraw | 0 | 0 | 1
Not completed — Subject/Guardian Decision to Withdraw | 0 | 0 | 12

BASELINE CHARACTERISTICS:
Population: Safety population: All patients who received any amount of rituximab or any vaccine.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab + Methotrexate (Group A) | Methotrexate (Group B) | Total
Number analyzed (Participants) | 68 | 32 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (9.60) | 49.7 (10.51) | 49.7 (9.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 25 | 76
  Male | 17 | 7 | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With a Positive Immune Response to Tetanus Toxoid Adsorbed Booster Vaccine
Description: The immune response to tetanus toxoid adsorbed booster vaccine was measured in serum samples immediately prior to and 4 weeks after vaccine administration. The tetanus antibody test was an ELISA that used tetanus toxoid as a capturing reagent and alkaline phosphatase-conjugated anti-human IgG (γ) for detection. For patients with pre-vaccination tetanus antibody titers < 0.1 IU/mL, a positive immune response was defined as an antibody titer ≥ 0.2 IU/mL. For patients with pre-vaccination tetanus antibody titers ≥ 0.1 IU/mL, a positive immune response to the booster immunization was defined as a 4-fold increase in antibody titer.
Time Frame: Week 24 to Week 28 for Group A and Day 1 to Week 4 for Group B
Population: Immune response per-protocol population: Group A - All patients randomized to Group A who received any rituximab infusion and any vaccine and had pre-vaccination and 4-week post-vaccination blood samples. Group B - All patients randomized to Group B who received any vaccine and had pre-vaccination and 4-week post-vaccination blood samples.
Measure: Number; unit: Percentage of patients
Arm/Group | Rituximab + Methotrexate (Group A) | Methotrexate (Group B)
Number analyzed (Participants) | 64 | 26
Percentage of patients | 39.1 | 42.3

2. Secondary Outcome: Percentage of Patients With a 2-fold Increase in Tetanus Antibody Titers or With Tetanus Antibody Titers ≥ 0.2 IU/mL in Response to Tetanus Toxoid Adsorbed Booster Vaccine
Description: The immune response to tetanus toxoid adsorbed booster vaccine was measured in serum samples immediately prior to and 4 weeks after vaccine administration. The tetanus antibody test was an ELISA that used tetanus toxoid as a capturing reagent and alkaline phosphatase-conjugated anti-human IgG (γ) for detection.
Time Frame: Week 24 to Week 28 for Group A and Day 1 to Week 4 for Group B
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Rituximab + Methotrexate (Group A) | Methotrexate (Group B)
Number analyzed (Participants) | 64 | 26
Percentage of patients | 54.7 | 61.5

3. Secondary Outcome: Percentage of Patients With a Positive Immune Response to Each of the 12 Anti-pneumococcal Antibody Serotypes in Response to the 23-valent Pneumococcal Polysaccharide Vaccine
Description: The immune response to each of the 12 anti-pneumococcal antibody serotypes was measured in serum samples immediately prior to and 4 weeks after vaccine administration. The pneumococcal antibody assay was a fluoroimmunoassay that used a Luminex Multiplex platform. Purified capsular polysaccharides isolated from 12 serotypes of S. pneumonia were covalently attached to microbeads and used as a capturing reagent. Phycoerythrin conjugated anti-human IgG was used for detection. A positive immune response against a serotype was defined as a 2-fold increase or an increase of > 1 μg/mL from pre-vaccination levels.
Time Frame: Week 28 to Week 32 for Group A and Week 4 to Week 8 for Group B
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Rituximab + Methotrexate (Group A) | Methotrexate (Group B)
Number analyzed (Participants) | 63 | 28
Percentage of patients
  Serotype 1-146 (1) | 12.7 | 42.9
  Serotype 3-146 (3) | 9.5 | 28.6
  Serotype 4-146 (4) | 12.7 | 60.7
  Serotype 6/26-146 (6B) | 38.1 | 60.7
  Serotype 8-146 (8) | 33.3 | 57.1
  Serotype 9-146 (9N) | 22.2 | 60.7
  Serotype 12-146 (12F) | 11.1 | 50.0
  Serotype 14-146 (14) | 30.2 | 60.7
  Serotype 19-146 (19F) | 25.4 | 53.6
  Serotype 23-146 (23F) | 20.6 | 35.7
  Serotype 51-146 (7F) | 25.4 | 60.7
  Serotype 56-146 (18C) | 20.6 | 57.1

4. Secondary Outcome: Percentage of Patients With a Positive Immune Response to at Least 50% (≥ 6 of 12) of the 12 Anti-pneumococcal Antibody Serotypes in Response to the 23-valent Pneumococcal Polysaccharide Vaccine
Description: as for outcome 3
Time Frame: Week 28 to Week 32 for Group A and Week 4 to Week 8 for Group B
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Rituximab + Methotrexate (Group A) | Methotrexate (Group B)
Number analyzed (Participants) | 63 | 28
Percentage of patients | 19.0 | 60.7

5. Secondary Outcome: Percentage of Patients With a Positive Immune Response to at Least k (for k = 1, 2, 3, 4, 5) of the 12 Anti-pneumococcal Antibody Serotypes in Response to the 23-valent Pneumococcal Polysaccharide Vaccine
Description: as for outcome 3
Time Frame: Week 28 to Week 32 for Group A and Week 4 to Week 8 for Group B
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Rituximab + Methotrexate (Group A) | Methotrexate (Group B)
Number analyzed (Participants) | 63 | 28
Percentage of patients
  1 serotype | 57.1 | 82.1
  2 serotypes | 42.9 | 82.1
  3 serotypes | 38.1 | 78.6
  4 serotypes | 33.3 | 75.0
  5 serotypes | 23.8 | 67.9

6. Secondary Outcome: Serum Level of Anti-tetanus Antibody Measured Immediately Prior to and 4 Weeks After Administration of a Tetanus Toxoid Adsorbed Booster Vaccine
Description: Anti-tetanus antibody was measured in serum samples immediately prior to and 4 weeks after administration of a tetanus toxoid adsorbed booster vaccine. The tetanus antibody test was an ELISA that used tetanus toxoid as a capturing reagent and alkaline phosphatase-conjugated anti-human IgG (γ) for detection.
Time Frame: Week 24 to Week 28 for Group A and Day 1 to Week 4 for Group B
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Rituximab + Methotrexate (Group A) | Methotrexate (Group B)
Number analyzed (Participants) | 64 | 26
IU/mL
  Pre-vaccination | 1.2 [0.88 to 1.69] | 1.0 [0.49 to 2.14]
  4 weeks post-vaccination | 4.0 [2.72 to 5.74] | 5.2 [2.25 to 12.00]

7. Secondary Outcome: Serum Level of Anti-pneumococcal Antibody Measured Immediately Prior to and 4 Weeks After Administration of a 23-valent Pneumococcal Polysaccharide Vaccine
Description: Anti-pneumococcal antibody was measured immediately prior to and 4 weeks after administration of a 23-valent pneumococcal polysaccharide vaccine. The pneumococcal antibody assay was a fluoroimmunoassay that used a Luminex Multiplex platform. Purified capsular polysaccharides isolated from 12 serotypes of S. pneumonia were covalently attached to microbeads and used as a capturing reagent. Phycoerythrin conjugated anti-human IgG was used for detection.
Time Frame: Week 28 to Week 32 for Group A and Week 4 to Week 8 for Group B
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Rituximab + Methotrexate (Group A) | Methotrexate (Group B)
Number analyzed (Participants) | 63 | 28
µg/mL
  Pre-vaccination | 0.8 [0.64 to 1.06] | 1.0 [0.68 to 1.47]
  4 weeks post-vaccination | 1.0 [0.76 to 1.37] | 2.3 [1.39 to 3.89]

8. Secondary Outcome: Serum Level of Anti-keyhole Limpet Hemocyanin Antibody Measured Immediately Prior to and 4 Weeks After the First Administration of Keyhole Limpet Hemocyanin
Description: Anti-keyhole limpet hemocyanin antibody was measured immediately prior to and 4 weeks after the first administration of keyhole limpet hemocyanin. The keyhole limpet hemocyanin antibody ELISA assay used keyhole limpet hemocyanin as the plate coat and anti-human IgG-horseradish peroxidase for detection.
Time Frame: Week 32 to Week 36 for Group A and Week 8 to Week 12 for Group B
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Rituximab + Methotrexate (Group A) | Methotrexate (Group B)
Number analyzed (Participants) | 64 | 27
IU/mL
  Pre-vaccination | 345.7 [312.25 to 382.76] | 388.0 [NA to NA] — The confidence interval could not be calculated as only 1 patient had an anti-body response above the lower limit of quantitation.
  4 weeks post-vaccination | 539.5 [461.54 to 630.61] | 1585.5 [1065.15 to 2360.17]

9. Secondary Outcome: Percentage of Patients Who Maintained a Positive Response to the C. Albicans Skin Test From Day 1 to Week 24 for Group A or From Day 1 to Week 12 for Group B
Description: Patients received an intradermal injection of C. albicans on the volar surface of the forearm on Day 1 and Week 24 for Group A or on Day 1 and Week 12 for Group B. Forty-eight to 72 hours after injection, patients were evaluated for a delayed-type hypersensitivity response by measuring the diameter of induration (palpable raised, hardened area of the forearm skin). A positive response to the C. albicans skin test was defined as at least 5 mm in diameter of induration.
Time Frame: Day 1 to Week 24 for Group A and Day 1 to Week 12 for Group B
Population: Skin test per-protocol population: Group A - All patients randomized to Group A who received any rituximab infusion, had Day 1 and Week 24 skin tests, and who provided complete diameter of induration readings. Group B - All patients randomized to Group B who had Day 1 and Week 12 skin tests and who provided complete diameter of induration readings.
Measure: Number; unit: Percentage of patients
Arm/Group | Rituximab + Methotrexate (Group A) | Methotrexate (Group B)
Number analyzed (Participants) | 64 | 28
Percentage of patients | 77.4 | 70.0

10. Secondary Outcome: Percentage of Patients in Group A With an Improvement of at Least 20%, 50%, or 70% in American College of Rheumatology (ACR) Score (ACR20/50/70) From Baseline at Week 24
Description: Improvement must be seen in tender and swollen joint counts (28 assessed joints) and in at least 3 of the following 5 parameters: Separate patient and physician assessments of patient disease activity in the previous 24 hours on a visual analog scale (VAS, the extreme left end of the line "no disease activity" [symptom-free and no arthritis symptoms] and the extreme right end "maximum disease activity"; patient assessment of pain in previous the 24 hours on a VAS (extreme left end of the line "no pain" and the extreme right end "unbearable pain"); Health Assessment Questionnaire-Disability Index (20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities, 0=without difficulty to 3=unable to do); and C reactive protein or, if missing, erythrocyte sedimentation rate.
Time Frame: Week 24
Population: Safety population: All patients who received any amount of rituximab or any vaccine. Since only limited efficacy data were collected in this study, the parameters necessary to calculate the ACR20/50/70 responses were only available for patients in Group A.
Measure: Number; unit: Percentage of patients
Arm/Group | Rituximab + Methotrexate (Group A)
Number analyzed (Participants) | 66
Percentage of patients
  ACR 20% | 36.4
  ACR 50% | 21.2
  ACR 70% | 4.5

ADVERSE EVENTS:
Time Frame: Adverse events were reported from Weeks 1-36 for Group A and Weeks 1-24 for Group B of the treatment period, Weeks 1-6 of the optional extension retreatment period, and Weeks 1-48 of the safety follow-up period (maximum of up to 90 weeks).
Description: Safety population: All patients who received any amount of rituximab or any vaccine.
Groups:
- Rituximab + Methotrexate (Group A) - Treatment Period: Patients received 2 intravenous infusions of rituximab 1000 mg, 14 days apart + methotrexate 10-25 mg/wk orally or subcutaneously during the Treatment Period.
- Methotrexate (Group B) - Treatment Period: Patients received methotrexate 10-25 mg/wk orally or subcutaneously during the Treatment Period.
- Group A - Optional Extension Re-treatment Period; Group B - Optional Extension Re-treatment Period: Patients who qualified for re-treatment received 2 intravenous infusions of rituximab 1000 mg, 14 days apart + methotrexate 10-25 mg/week orally or subcutaneously. Patients received methylprednisolone 100 mg intravenously before each infusion of rituximab.
- Group A - Safety Follow-up Period; Group B - Safety Follow-up Period: Patients received no treatment during the Safety Follow-up Period.
Arm/Group | Rituximab + Methotrexate (Group A) - Treatment Period | Methotrexate (Group B) - Treatment Period | Group A - Optional Extension Re-treatment Period | Group B - Optional Extension Re-treatment Period | Group A - Safety Follow-up Period | Group B - Safety Follow-up Period
Serious Adverse Events (participants affected / at risk) | 3/68 | 2/32 | 2/52 | 2/26 | 3/68 | 1/32
Other Adverse Events (participants affected / at risk) | 51/68 | 19/32 | 7/52 | 13/26 | 19/68 | 11/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + Methotrexate (Group A) - Treatment Period (N=68) | Methotrexate (Group B) - Treatment Period (N=32) | Group A - Optional Extension Re-treatment Period (N=52) | Group B - Optional Extension Re-treatment Period (N=26) | Group A - Safety Follow-up Period (N=68) | Group B - Safety Follow-up Period (N=32)
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hip fracture (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Amaurosis fugax (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + Methotrexate (Group A) - Treatment Period (N=68) | Methotrexate (Group B) - Treatment Period (N=32) | Group A - Optional Extension Re-treatment Period (N=52) | Group B - Optional Extension Re-treatment Period (N=26) | Group A - Safety Follow-up Period (N=68) | Group B - Safety Follow-up Period (N=32)
Nausea (Gastrointestinal disorders) | 7 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 7 | 2 | 1 | 4 | 8 | 6
Sinusitis (Infections and infestations) | 5 | 0 | 2 | 3 | 7 | 2
Influenza (Infections and infestations) | 5 | 1 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 12 | 0 | 0 | 2 | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 1 | 2 | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 9 | 3 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 2 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 0 | 3 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 6 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 3
Ear pruritus (Ear and labyrinth disorders) | 1 | 3 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 4 | 0 | 0 | 2 | 0 | 0
Feeling hot (General disorders) | 2 | 2 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 4 | 0 | 0 | 0 | 0 | 0
Genital herpes (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 0 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 3 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 4 | 2 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 5 | 1 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 4 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.